CLINICAL TRIAL: NCT03949777
Title: Validation of Aer-O-Scope Colonoscope System Cecal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI View Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1056CLD
Record Dates: First submitted 2019-04-28; First posted 2019-05-14 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-08

CONDITIONS: Colonic Polyp; Colonic Neoplasms; Colonic Diseases; Colon Adenoma; Colon Disease; Colon Adenocarcinoma; Colon Cancer
Keywords: screening-colonoscopy; diagnostic-colonoscopy; surveillance-colonoscopy
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms; Colonic Diseases

STUDY DESIGN:
Intervention Model Description: A single group of subjects will undergo diagnostic, screening or surveillance colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Cohort (Experimental): 61 subjects will undergo colonoscopy
  Interventions: Device: Aer-O-Scope Colonoscopy

INTERVENTIONS:
Device: Aer-O-Scope Colonoscopy — resection or biopsy of colonic abnormalities for histopathalogical evaluation
  Other Names: therapeutic intervention - polyp resection

SUMMARY:
61 subjects (male or female) between the ages of 45 and 75 will undergo colonoscopy. The primary outcome is Cecal Intubation

DETAILED DESCRIPTION:
This will be a prospective single-center non-blinded clinical investigation. Each subject will undergo a colonoscopy to the cecum with the Aer-O-Scope Colonoscope System. All pathologies found will be removed. No control group is necessary as the main objective is to reach the cecum. Either the cecum is intubated or it is not. This is true for all colonoscopy procedures.

Up to the first ten (10) cases for each physician will be system operation training cases.

The primary endpoint of cecal intubation was chosen as this measure is the first quality objective when evaluating colonoscopy quality indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is indicated for screening, diagnostic (minor complaints such as rectal bleeding or minor abdominal pain) or surveillance colonoscopy
2. Subject willing to undergo colon preparation bowel cleansing
3. Subject between the ages of 45 and 75 (patients between the ages of 45 and 50 must have a family history of a first degree relative with onset of colon cancer before the age of 60).
4. Subject is able to understand and willing to sign informed consent form

Exclusion Criteria:

1. Personal history of colorectal neoplasia including familial adenomatous polyposis or hereditary nonpolyposis, colon cancer (HNPCC).
2. Diagnosis of active (flaring) inflammatory bowel disease (active ulcerative colitis or Crohn's colitis), bowel obstruction, or acute diverticulitis, or known severe diverticulosis, fecal incontinence or any known large-bowel disease that would require a predetermined therapeutic colonoscopy (non-screening, non-diagnostic or non-surveillance cases)
3. Severe gastrointestinal tract-related symptoms, or complaints, suggesting performance of a pre-determined therapeutic colonoscopy (non-screening, non-diagnostic or non-surveillance cases)
4. History of colonic resection
5. Clinically significant cardiovascular or pulmonary disease.
6. Cancer or other life threatening disease or significant chronic condition that puts the subject at risk.
7. Blood-clotting disorders and/or current anticoagulant therapy (Subjects taking up to 100mg aspirin for prophylactic treatment are acceptable for this study)
8. Pregnancy
9. Previous radiation therapy to the abdomen
10. Morbid Obesity (BMI > 40 kg/m2)
11. Drug abuse or alcoholism
12. Subject is bed-ridden and/or unable to adequately communicate
13. Subject is under custodial care
14. Subject has a history of psychiatric disorders which would prevent compliance with study instructions
15. Participation in a clinical study within the previous 30 days

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Aer-O-Scope Validation of Cecal Intubation | 30 minutes
  The number of subjects for which cecal intubation will be achieved using the Aer-O-Scope Disposable Colonoscope

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Gluck, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared